CLINICAL TRIAL: NCT07001683
Title: The Effect of Virtual Reality Respiratory and Physical Exercises on Self-Efficacy and Quality of Life in COPD Patients
Brief Title: The Effect of Virtual Reality on Self-Efficacy and Quality of Life in COPD Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emrah Ay (Other)
Collaborators: Ataturk University (Other); Prof. Dr. Mağfiret Kaşıkçı (Unknown)
Responsible Party: Sponsor-Investigator, Emrah Ay, research assistant, Ataturk University
Organization: Ataturk University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: AtaturkU-EAy-001
Record Dates: First submitted 2023-09-13; First posted 2025-06-03 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-05

CONDITIONS: Nursing Caries; Copd; Cough; Quality of Life; Self Efficacy
Keywords: breathing exercise,; COPD; PHYSICAL EXERCISE; quality of life; virtual reality; self efficacy
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Cough; Motor Activity

STUDY DESIGN:
Intervention Model Description: Population and Sample of the Research The population of this research consisted of individuals receiving inpatient treatment at the Chest Diseases Clinic of Atatürk University Research and Application Center between December 2021 and June 2022, and patients with COPD who applied to the outpatient clinic.
  In the study, post-test data could not be collected due to the death of two patients in the control group, and the control group was terminated with 30 patients, and the study was completed with 62 patients in total, 32 experimental and 30 control. Reporting of the study was done according to the CONSORT (Consolidated Standards of Reporting Trials) randomized controlled trials guide. The patients were randomly divided into 2 groups: experimental group n=32 and control group n=32, by block randomization method using the "random.org" website. The Randomization Scheme according to the CONSORT 2018 diagram.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EXPERIMENTAL GROUP PATIENT (Experimental): Through the video content, patients are given practical breathing and physical exercises through a mentor in a virtual environment. Before the videos were shown to the patients, detailed information was given about how to use the glasses, what to do and the video content, and they were asked to apply the visual and verbal commands given on the screen. Virtual reality application was performed outside the treatment and examination hours when the patient felt well, at a time when his vital signs and oxygen saturation were within normal limits. The first virtual reality application was made in the hospital and the patients were observed. Patients who could not perform the exercises were completed the exercises according to the step-by-step instructions given by the researcher as support. Patients who could perform the exercises without any problems were loaned glasses for virtual reality applications and were asked to do the exercises on their own at home for 6 weeks.
  Interventions: Device: VR SHINECON VIRTUAL REALITY GLASES
- CONTROL GROUP PATIENT(unattended) (Active Comparator): Control Group (unattended) The patients were interviewed face to face and completed the questionnaires, then they were told to use their medications as prescribed by the doctors, and they were interviewed again after 6 weeks and the forms were filled out. No intervention was applied to the patients in the control group. Interviews lasted approximately 30 minutes for each patient.
  Interventions: Device: VR SHINECON VIRTUAL REALITY GLASES

INTERVENTIONS:
Device: VR SHINECON VIRTUAL REALITY GLASES — Unity program; It is a game engine that is used for the development of 2D, 3D, virtual reality and augmented reality applications and also has mobile support. 3D objects and animations necessary to develop the application have been prepared. These objects and animations; It was developed in the Autodesk 3ds Max program, where 3D modeling and animations are made.
  The virtual reality aspect of the application is integrated into the Google VR SDK (Google Virtual Reality Software Development Kit). Interactions in the virtual environment and 360° viewing operations in the virtual world are provided through this Google VR SDK. The development process was completed by writing application codes in C#, one of the languages supported by the Unity program, using the methods included in the SDK.
  Other Names: Software Developed for Virtual Reality Module

SUMMARY:
Introduction: Chronic obstructive pulmonary disease (COPD) is a serious chronic disease worldwide with significant adverse effects on patients' quality of life, family economic burden and social health care burden. The aim of this study was to investigate the effects of breathing and cough exercises performed with virtual reality technology on quality of life and self-efficacy in COPD patients.

Methods: The study was conducted as a pre-test post-test randomised controlled experimental study. The study included 64 patients with COPD, randomly assigned to receive virtual reality-based breathing and exercises (experimental group n=32) and patients receiving routine clinical treatment (control group, n=32). Interventions were conducted three times a week for 6 weeks. Google VR SDK (Google Virtual Reality Software Development Kit) was used for the training of the experimental group. In the evaluation of the data; mean, number, percentage distributions, dependent and independent groups t-test analysis methods were used.

DETAILED DESCRIPTION:
Research Type This research; It was planned as a randomized controlled study to determine the effects of breathing and physical exercises performed with virtual reality on self-efficacy and quality of life in COPD patients.

Location and Characteristics of the Research Research data was collected between December 2021 and June 2022 at the Atatürk University Research and Application Center Chest Diseases clinic and polyclinic.

Atatürk University Research and Application Center Chest Diseases Clinic has 36 beds and approximately 60 patients are admitted per month, and patients stay in the clinic for an average of 5-15 days. The clinic operates 24 hours a day, 7 days a week, throughout the year. In the clinic, 2 doctors, 2 nurses, 1 secretary and 2 assistant staff work in the 08:00-16:00 shift, and 1 doctor, 1 nurse and 1 assistant work in the 16:00-24:00 shift. 00-08:00 shift. personnel are on duty. The chest diseases outpatient clinic serves patients on weekdays and has two examination rooms in total. There are two separate rooms in the chest clinic where respiratory function tests are performed, and these test measurements are made by nurses.

Population and Sample of the Research The population of this research consisted of individuals receiving inpatient treatment at the Atatürk University Research and Application Center Chest Diseases Clinic between December 2021 and June 2022 and COPD patients who applied to the outpatient clinic.

A priori power analysis was performed to determine the number of samples. Cohen's standard effect sizes were used as the reference method in the power analysis. In the power analysis, there must be at least 26 people in both groups to reach 80% power with a p<0.05 significance level, a high effect size and a 95% confidence interval in two groups with pre-test and post-test. Scale. It was determined that a total of 52 participants were needed. 123 However, considering that there would be data loss, 32 patients were included in both groups.

Research Inclusion Criteria

Those diagnosed with COPD as a result of pulmonary function tests (FEV1/FVC < 70%) Does not have any psychiatric problems, Having COPD group B or C for at least three months according to the GOLD (2019) classification, Those who have not received breathing exercise training before and have not participated in any rehabilitation program, Residing in the city center where the research is conducted, Enough to understand the questions Does not have any vision or hearing problems, Open to communication and collaboration, Patients who volunteered to participate in the study were included.

ELIGIBILITY:
Inclusion Criteria:

* Those diagnosed with COPD as a result of pulmonary function tests (FEV1/FVC < 70%)
* Having no psychiatric problems,
* Having COPD group B or C for at least three months according to the GOLD (2019) classification,
* Those who have not received breathing exercise training before and have not participated in a rehabilitation program,
* Living in the city center where the study is carried out,
* Sufficient to understand the questions,
* Having no problems with vision or hearing,
* Open to communication and collaboration,
* Patients who volunteered to participate in the study were included.

Exclusion Criteria:

* being under 18 years old unwilling to cooperate not diagnosed with COPD

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2023-01-01 (Actual); Study Completion 2023-02-10 (Actual)

PRIMARY OUTCOMES:
COPD Assessment Test (CAT | before application
  COPD Assessment Test (CAT) mean score decreases, and patients' health status improves with the decrease in CAT scores

SECONDARY OUTCOMES:
COPD Assessment Test (CAT | 6 weeks later
  COPD Assessment Test (CAT) mean score decreases, and patients' health status improves with the decrease in CAT scores.

CONTACTS AND LOCATIONS:
Overall Officials: MAĞFİRET KAŞIKÇI, Study Director — Advısor
Locations (1):
- Atatürk Üniversitesi, Erzurum, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Agusti A, Vogelmeier C, Faner R. COPD 2020: changes and challenges. Am J Physiol Lung Cell Mol Physiol. 2020 Nov 1;319(5):L879-L883. doi: 10.1152/ajplung.00429.2020. Epub 2020 Sep 23. No abstract available. PMID 32964724
- [Background] Kara M, Asti T. Effect of education on self-efficacy of Turkish patients with chronic obstructive pulmonary disease. Patient Educ Couns. 2004 Oct;55(1):114-20. doi: 10.1016/j.pec.2003.08.006. PMID 15476998
- [Background] Xie X, Fan J, Chen H, Zhu L, Wan T, Zhou J, Fan D, Hu X. Virtual Reality Technology Combined with Comprehensive Pulmonary Rehabilitation on Patients with Stable Chronic Obstructive Pulmonary Disease. J Healthc Eng. 2021 Aug 2;2021:9987200. doi: 10.1155/2021/9987200. eCollection 2021. PMID 34394902
- See also: goldcopd — http://goldcopd.org/wp-content/uploads/2020/11/GOLD-REPORT-2021-v1.1-25Nov20_WMV.pdf